CLINICAL TRIAL: NCT02162173
Title: Diagnostic Values of Dual Focus Narrow Band Imaging and Probe-based Confocal Laser Endomicroscopy in FAP Related Duodenal Adenoma
Brief Title: Dual Focus NBI and pCLE in FAP Related Duodenal Adenoma
Acronym: PIVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Doctor, King Chulalongkorn Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP007
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Complication of Diagnostic Procedure; Adverse Effect of Diagnostic Agents, Subsequent Encounter
Keywords: Familial adenomatous polyposis syndrome; Non-ampullary polyp; Ampullary polyp; Narrow band imaging endoscopy; Confocal laser endomicroscopy
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Endoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopy (Experimental): All patients underwent the same endoscopy.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopist performed white light endoscopy for polyp detection, then switch to dual focus NBI for characterization. Then probe-based confocal laser endomicroscopy was applied for characterization by another endoscopist independently and finally biopsy.
  Other Names: White light endoscopy; dual focus NBI endoscopy; probe-based confocal laser endomicroscopy; biopsy

SUMMARY:
Background: Familial adenomatous polyposis (FAP) patients are at risk to develop periampullary and non-ampullary adenoma. Either a routine biopsy or an endoscopic removal of the lesion is generally required to identify the presence of adenoma. However, the risk of tissue sampling from the ampulla is high and non-ampullary polyps are sometimes numerous, therefore resecting all the lesions is time consuming. To support the PIVI (Preservation and Incorporation of Valuable endoscopic Innovations) initiative, a real-time diagnosis with NPV≥ 90% is required.

Objective: To evaluate the diagnostic values of duodenal adenoma by dual focus NBI (dNBI) and probe-based confocal endomicroscopy (pCLE) in FAP patients.

Design: Diagnostic study.

Setting: Single tertiary-care referral center.

Patients: Twenty-six patients with previously diagnosed with FAP.

Intervention: Surveillance EGD with dNBI and pCLE. A real time adenoma reading was done by two different endoscopists for each of the technique. Histology from the matched lesion was used as the gold standard.

Main outcome measurements: Sensitivity, specificity, positive predictive value (PPV), and accuracy. With the threshold for negative predictive value (NPV) ≥ 90%

DETAILED DESCRIPTION:
Endoscopic procedure and criteria for adenoma diagnosis

* The endoscopic diagnostic criteria to distinguish between adenoma and non-adenoma were adopted from the previous studies by Uchiyama Y et al. in 2006. A real time adenoma diagnosis was made by the two independent endoscopists (BI and RP) who are experienced in dNBI and pCLE readings. Before entering into the study, they have experienced in reviewing the images obtained by dNBI and pCLE and published the related results elsewhere.
* During the study period, all 26 patients underwent the procedure under conscious sedation with intravenous midazolam and meperidine. Ten milligrams of hyoscine was given before the procedure to decrease intestinal peristalsis. At the beginning of the procedure, the first endoscopist (BI) used an end-viewing HWE attached with an endoscopic cap to examine the 1st and 2nd part of duodenum. The cap was used to facilitate a proper enface view of the ampulla and surrounding area. All applicable ampullary and non-ampullary (duodenal) polyps that larger than 1 millimeter would be recruited in this study. Then dNBI mode was switched on for a real-time diagnosis by the first endoscopist (BI). Subsequently, the second endoscopist (RP) who blinded to the NBI reading would be called from another room to perform pCLE examination. Two and a half milliliters of 10% fluorescein (Novartis Pharmaceutical Corporation, Bangkok, Thailand) was injected during pCLE evaluation. When there were more than one non-ampulary lesions, the first endoscopist only navigated the lesions to study under pCLE to the second endoscopist without telling the result of dNBI reading. Then, the matched polypectomy or biopsy was performed by the second endoscopist. The duration of the entire procedure and all complications related to the procedures were recorded.

Histological assessment - All polypectomy and biopsy specimens were immersed in formalin and sent for histological examination. The specimens were stained with hematoxylin and eosin (H&E) and reviewed by an experienced GI pathologist (NW) blinded to the endoscopic diagnosis. The definite diagnosis was based on the Vienna classification for differentiation between adenoma and non-adenoma.

Statistical Analysis

-By using histology as the gold standard, the diagnostic values of dNBI and pCLE for ampullary and non-ampullary polyp interpretation were assessed for sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy. According to PIVI recommendation for colonic adenoma diagnosis20, we used the 90% NPV readings as our cut off. For numerical variables, the results were expressed as a mean ± SD, whereas other quantitative variables are expressed as percentages. SPSS version 17.0 (SPSS (Thailand) Co., Ltd., Bangkok, Thailand) for Windows systems was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with a history of FAP
* Patients who able to provide a written informed consent.

Exclusion Criteria:

* Evidence of coagulopathy (INR ≥ 1.5 and/or platelet < 80,000)
* Other bleeding tendency precluding biopsy
* Pregnancy
* allergy to fluorescein sodium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
duodenal adenoma diagnosis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Patumwan, Bangkok, Thailand

REFERENCES:
- [Derived] Pittayanon R, Rerknimitr R, Imraporn B, Wisedopas N, Kullavanijaya P. Diagnostic values of dual focus narrow band imaging and probe-based confocal laser endomicroscopy in FAP-related duodenal adenoma. Endosc Int Open. 2015 Oct;3(5):E450-5. doi: 10.1055/s-0034-1392235. Epub 2015 Jun 23. PMID 26528500